CLINICAL TRIAL: NCT07109947
Title: Comparison Between the Use of Aromatase Inhibitor Before Misoprostol and Use of Misoprostol Alone in Medical Termination of Miscarriage
Brief Title: Use of Aromatase Inhibitor Before Misoprostol in Medical Termination of Miscarriage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Arwa Ashraf Saeed, Demonstrator at Obstetrics and Gynecology, Faculty of medicine, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arwa Ashraf
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: letrozole and Misoprostol (Active Comparator): About 35 pregnant women will receive aromatase inhibitor (letrozole) 2.5 mg tablet three times daily for 3 days followed by two doses of 400 micrograms of misoprostol administered vaginally on the 4th day of enrolment (two 200-μg tablets spaced 4 hours apart).
  Interventions: Drug: Letrozole 2.5mg
- Group B: Misoprostol (Active Comparator): About 35 pregnant women will receive two doses of 400 µg of vaginal misoprostol (two 200-μg tablets spaced 4 hours apart).
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Letrozole 2.5mg — to determine the effect of Letrozole as a premedication before misoprostol treatment used to induce missed miscarriage.
  Other Names: Misoprestol

SUMMARY:
Abortion is one of the most common complications of pregnancy. Missed abortion is a type of abortions, occurs in 15%-20% of clinically diagnosed pregnancies and is defined as the retention of pregnancy products in the uterus for several days or weeks after death of the fetus.

DETAILED DESCRIPTION:
Various medical and surgical methods have been used to manage missed abortions. Surgical methods include dilatation and curettage, and vacuum aspiration. Because these methods are expensive and involve anesthesia, however, medical methods are generally preferred over surgical methods for abortion.

Medical approaches include misoprostol which is a prostaglandin that causes myometrial contractions, cervical softening and dilatation. It is used to induce abortion and labor and to treat atonic postpartum hemorrhage and peptic ulcers.

It has the advantage of being cost-effective and stable with a low rate of side effects which has led to it being included in the World Health Organization list of essential medications (2014). Misoprostol is licensed for use to induce miscarriage in Egypt. It has not been licensed to induce labor or miscarriage in certain countries such as Germany, but it is used off-label to induce labor in the UK.

Usage of Misoprostol alone has a success rate of between 65 and 93% especially in the early stages of pregnancy. It can also use in combination with other medications such as mifepristone and methotrexate to increase the success rate.

Most studies have examined the effect of letrozole plus misoprostol on the abortion of live embryos .Given the significance of specifying an effective and safe method for termination of abortion and the specific features of letrozole, such as its safety, cost-effectiveness, and availability.

ELIGIBILITY:
Inclusion Criteria:

* Missed or anembryonic pregnancy.
* Gestational age from 4 weeks to 26 weeks of pregnancy (confirmed by ultrasound scanning on first day of admittance).
* Hemoglobin level more than 9g/l.
* Closed cervix.
* No product of conception in the cervical canal.

Exclusion Criteria:

* Previous attempt to terminate the pregnancy.
* Molar pregnancy
* Abnormal uterine lesions such as fibroids or congenital mal formations.
* Pregnancy despite of intrauterine contraceptive device.
* Medical disorders as cardiac, renal or hemorrhagic diseases.
* BMI more than 35 kg/m2.
* Known hypersensitivity to any of the medication used.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Miscarriage Achievement | 10 days
  The induction-to-abortion interval in each group

CONTACTS AND LOCATIONS:
Overall Officials: Hani Ahmed Farouk, Assist.Prof., Study Chair — Obstetrics and Gynecology,Faculty of Medicine,Aswan University
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided